CLINICAL TRIAL: NCT02644226
Title: Retrospective Investigation of Perioperative Upper Airway Complications After Anesthesia Using Supraglottic Airway Devices in Children: Comparison of Desflurane and Sevoflurane
Brief Title: Laryngeal Mask Airway (LMA) Complication in Children
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, AH-YOUNG OH, Dr., Seoul National University Bundang Hospital
Other Study IDs: B-1407/258-117
Record Dates: First submitted 2015-12-23; First posted 2015-12-31 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Laryngeal Mask Airway
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sevoflurane: The investigators retrospectively reviewed and analyzed the electrical medical records of consecutive children aged 1 to 15 years who underwent general anesthesia under supraglottic airways using sevoflurane as maintenance agents.
  Interventions: Other: Sevoflurane
- Desflurane: The investigators retrospectively reviewed and analyzed the electrical medical records of consecutive children aged 1 to 15 years who underwent general anesthesia under supraglottic airways using desflurane as maintenance agents.
  Interventions: Other: Desflurane

INTERVENTIONS:
Other: Sevoflurane — The investigators retrospectively reviewed and analyzed the electrical medical records of consecutive children aged 1 to 15 years who underwent general anesthesia under supraglottic airways using sevoflurane as maintenance agents.
  Groups: Sevoflurane
Other: Desflurane — The investigators retrospectively reviewed and analyzed the electrical medical records of consecutive children aged 1 to 15 years who underwent general anesthesia under supraglottic airways using desflurane as maintenance agents.
  Groups: Desflurane

SUMMARY:
Desflurane is known to be the most pungent of the currently used volatile anesthetics. The investigators tried to find out if desflurane increases the incidence of perioperative upper airway complications in infants and children undergoing general anesthesia using supraglottic airways compared to sevoflurane.

DETAILED DESCRIPTION:
The investigators retrospectively reviewed and analyzed the electrical medical records of consecutive children aged 1 to 15 years who underwent general anesthesia under supraglottic airways using sevoflurane or desflurane as maintenance agents.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to 15 years who underwent general anesthesia under supraglottic airways using sevoflurane or desflurane as maintenance agents

Exclusion Criteria:

* Tracheal intubation

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1 to 15 years who underwent general anesthesia under supraglottic airways using sevoflurane or desflurane as maintenance agents in Seoul National University Bundang Hospital between June 2013 and June 2015.
Sampling Method: Non-Probability Sample
Enrollment: 3528 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of Laryngospasm | intraoperative
Occurrence of Cough | intraoperative
Occurrence of desaturation | intraoperative

SECONDARY OUTCOMES:
Occurrence of Laryngospasm | through study completion, an average of 1 day
Occurrence of desaturation | through study completion, an average of 1 day
Occurrence of Cough | through study completion, an average of 1 day

IPD SHARING:
Plan to Share IPD: No